CLINICAL TRIAL: NCT06422169
Title: Interventistic Monocentric Pre-market Clinical Investigation on the Use of Medical Device "ArToFILL" in Subjects With Mild-moderate Osteoarticular Pain
Brief Title: Interventistic Clinical Investigation on the Use of Medical Device in Subjects With Mild-moderate Osteoarticular Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PromoPharma spa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARTO/09/2023
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artofill (Experimental): One vial for intra-articular infiltration every 7 days, for three consecutive weeks. After the injection it is necessary to keep the infiltrated joint at rest for at least 24 hours. In addition, as with all invasive joint treatments, the patient is advised to avoid any physical activity 2-3 days after the injection. Do not repeat the treatment before 7 days from the previous one.
  Interventions: Device: ArToFILL

INTERVENTIONS:
Device: ArToFILL — ArToFILL is an injectable medical device (class III) intended for use as a temporary filler in joints. It is a sterile, non-pyrogenic, colorless and transparent hyaluronic acid gel of non-animal origin. ArToFILL is a hydrogel consisting of a mixture of two different molecular weights of hyaluronic acid, for a total HA concentration of 2.7 %.

SUMMARY:
Evaluation of the performance and safety of ArToFILL in subjects with mild to moderate osteoarticular pain

DETAILED DESCRIPTION:
Monocenter, prospective, open label, interventional clinical investigation evaluating the performance and safety of 3 intra-articular injections of ArToFILL for the treatment of mild-moderate osteoarticular pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient (males and females) aged between 18 and 84 years (limits included);
* Patient able to understand the nature and purpose of the study, including possible risks and side effects;
* Patient able to provide written Informed Consent, in accordance with good clinical practice and current legislation;
* Pain ≥ 40 mm on the VAS score in the target knee for at least 2 months;
* Patient with knee osteoarthritis assessed radiographically, grade 1 to 3 according to the Kellgren-Lawrence scale (K-L);
* Body Mass Index (BMI) ≤ 35;
* Patient who will benefit from this treatment;
* Patient available for the entire study period;
* Patient able to cooperate and meet the requirements of the clinical investigation plan.

Exclusion Criteria:

* Patient with knee osteoarthritis, assessed radiographically, grade 4 by the K-L scale;
* Patient presenting ongoing inflammation/infection at the level of the joint being investigated;
* Patient with abundant intra-articular effusion;
* Patient with symptoms of viral or bacterial infections or similar;
* Patient with insertion point of the joint infected or in the presence of a skin disease;
* Simultaneous treatment with disinfectants containing quaternary ammonium salts or chlorhexidine;
* Patient with known or potential allergy or hypersensitivity and/or history of allergic reactions to one of the components of the medical device;
* Concomitant treatments with thrombolytic or anticoagulant therapies, for less than 2 weeks prior to the screening visit;
* Intra-articular treatments carried out in the last 3 months (9 months if with products containing hyaluronic acid) of the target joint;
* Topical treatments of the target joint in progress or performed within 1 week of the screening visit;
* Taking NSAIDs and/or paracetamol as rescue treatment for more than two consecutive days;
* Surgical interventions of prosthetic replacement in the target joint;
* Physiotherapy and instrumental physical therapy treatments for the target joint performed in the last 2 weeks prior to the screening visit, and during the study period;
* Participation in another clinical trial within 60 days prior to the screening visit;
* Evidence of severe or uncontrolled systemic disease or any other significant disorder (e.g. haemophilia, bleeding disorders etc.); which do not allow participation in the study or could compromise the results.
* Patients who are pregnant or breastfeeding;
* Subject unable to follow clinical investigation procedures and follow-up visits;
* Any other medical condition which could influence participation in the clinical investigation or compromise its results.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-03-08 (Estimated); Study Completion 2025-05-08 (Estimated)

PRIMARY OUTCOMES:
Reduction ≥ of 15 points on VAS scale, at the Study Termination Visit compared to baseline | Up to 180 days
  Assessment of pain reduction using the visual analogue scale (VAS) ranging from 0 to 100 mm (where 0 = absent and 100 = strongest pain)

SECONDARY OUTCOMES:
Clinical improvement assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Up to 180 days
  Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. The total score is the result of the sum of 3 groups of questions with 5 possible answers (between 0 and 4, where 0=none and 4=extreme) for the self-assessment of:
  * pain:five questions (score from 0 to 20);
  * joint stiffness: two questions (score from 0 to 8);
  * functional limitations: 17 questions (score from 0 to 68).
Improved range of motion (ROM) of the knee joint | Up to 180 days
  The variation of the ROM joint excursion used for the analysis of the joint excursion (flexion-extension), will be calculated as the difference between maximum width and minimum width of the angular profile on the basis of the following formula: ROMα = max (α) - min (α) (flexion-extension)

OTHER OUTCOMES:
Evaluation of the safety and tolerability of treatment of medical device. | 180 days
  Investigator Global Assessment of Safety (IGAS): using the 4- point scale:1= very good safety, 2 =good safety, 3 = moderate safety and 4 = poor safety.
  Counting the number of files used for the patient confirmed by the number of traceability labels detached and kept by the Investigator
Evaluation of the safety and tolerability of treatment of medical device. | Up to 180 days
  Evaluation of reported adverse effects/incidents, monitoring of concomitant treatments, and the possible intake of rescue medication, assessment of patient compliance with the medical device in the study,

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vecchio, Principal Investigator — Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco", P.O. "G. Rodolico"
Locations (1):
- U.O. Recupero e riabilitazione funzionale P.O. "G.Rodolico", Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco", Catania, Italy

IPD SHARING:
Plan to Share IPD: No